CLINICAL TRIAL: NCT00496873
Title: A Single-Center, Open-Label Study to Evaluate the Safety and Efficacy of Nipent, Cytoxan, and Rituxan ("PCR") in the Treatment of Previously Untreated and Treated, Stage III or IV, Low-Grade B-Cell Non-Hodgkin's Lymphoma or Bulky Lymphoma
Brief Title: Evaluation of the Safety and Efficacy of Nipent, Cytoxan, and Rituxan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Pharmatech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0818; NCI-2010-00635 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2016-08-23 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Lymphoma
Keywords: Non-Hodgkin's Lymphoma; NHL; Lymphoma; B-cell chronic lymphocytic leukemia; SLL; Small Lymphocytic Lymphoma; Lymphoplasmacytic lymphoma/immunocytoma; Follicular lymphoma; Extranodal marginal zone B-cell lymphoma of MALT type; Nodal marginal zone B-cell lymphoma; Chronic Lymphocytic Leukemia; CLL; Bulky Lymphoma; Nipent; Cytoxan; Rituxan; Cyclophosphamide; Rituximab; Pentostatin
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular | interventions — Cyclophosphamide; Pentostatin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cytoxan + Rituxan + Nipent (Experimental): Cytoxan 600 mg/m^2 on Day 1 of 21-day cycle. Rituxan 375 mg/m^2 on Day 1 of 21 Day Cycle. Nipent 4 mg/m^2 on Day 1 of 21 Day Cycle.
  Interventions: Drug: Cytoxan; Drug: Nipent; Drug: Rituxan

INTERVENTIONS:
Drug: Cytoxan — 600 mg/m^2 on Day 1 of 21-day cycle.
  Other Names: Cyclophosphamide; Neosar
Drug: Nipent — 4 mg/m^2 on Day 1 of 21 Day Cycle.
  Other Names: Pentostatin; Deoxycoformycin; DCF
Drug: Rituxan — 375 mg/m^2 on Day 1 of 21 Day Cycle.
  Other Names: Rituximab

SUMMARY:
The goal of the clinical research study is to learn if treatment with a combination of three drugs, Cytoxan (cyclophosphamide), Rituxan (rituximab) and Nipent (pentostatin), will help to control the disease in patients with previously untreated non-Hodgkin's lymphoma, CLL, or bulky lymphoma. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
All of the drugs [Cytoxan (cyclophosphamide), Rituxan (rituximab) and Nipent (pentostatin)] in this study are commonly used in the treatment of this cancer. However, using these drugs in combination is investigational.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam. You will have blood collected (around 2-3 tablespoons) for routine tests. You will have a chest x-ray and CT scans of the chest, abdomen (stomach), and pelvis (waist area). Tumors will be measured using x-rays. You will have a sample of bone marrow collected. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. If your doctor feels it is necessary, you may also have lymph node biopsy samples taken for special tests. Women who are able to have children must have a negative blood or urine pregnancy test.

During treatment you will be given a combination of three drugs in a 21 day (3 weeks) cycle. All drugs will be given through a needle in a vein over 4-6 hours. You will receive pentostatin first, then rituximab, and lastly cyclophosphamide. For each treatment cycle cyclophosphamide, rituximab, and pentostatin will be given on Day 1, followed by 20 days of rest.

During treatment, you will have around 2-3 tablespoons of blood collected at least once a week for routine tests. You will also provide a urine sample for routine urine tests. Depending on how the disease responds, treatment may be stopped after 3, 6, or 9 cycles. You will be taken off treatment if your disease gets worse. If your treatment is delayed for more than 2 weeks due to any side effect related to the treatment or for more than 3 weeks for any reason, you will be taken off of this study. If your doctor feels that you are having serious or intolerable side effects that are not improved by standard supportive care methods (such as medicine to control nausea or a transfusion to treat anemia) you will be taken off of this study.

After Cycles 3, 6, and 9, tumors will be measured using x-rays or other scans (CT or MRI). Bone marrow samples will be taken if they are needed to find out if the drug combination is working to control your disease.

The maximum number of cycles that you can receive is 9. If you wish to continue using this drug treatment, and it is beneficial to do so, you may continue to receive these drugs. However, these drugs are commercially available, so you will be financially responsible for the cost of these drugs.

After you receive the last cycle of chemotherapy, your doctor will decide your schedule of follow-up exams. You will have follow-up exams every 3 months for one year, every 6 months for 2nd year, then once after 1 year. During these exams, you will have a chest x-ray and CT scans of the chest, abdomen (stomach), and pelvis (waist area). You will also have blood collected (2-3 tablespoons) for routine tests.

This is an investigational study. All of the study drugs are approved by the FDA for cancer treatment and are commercially available. However, the use of the drugs in combination is investigational. Up to 100 patients will take part in this study. All enrolled will be at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven, stage III or IV, low-grade B-cell NHL, as defined by the updated WHO modification of the REAL classification for peripheral B-cell neoplasms: B-cell chronic lymphocytic leukemia/small lymphocytic lymphoma; Lymphoplasmacytic lymphoma/immunocytoma; Follicular lymphoma; Extranodal marginal zone B-cell lymphoma of MALT type; Nodal marginal zone B-cell lymphoma (+/- monocytoid B-cells); Lymphoma with primarily bone marrow-only disease are considered eligible
2. Bulky lymphoma or Stage II disease requiring chemotherapy will be considered for enrollment with documented Sponsor Investigator approval prior to registration.
3. CT or MRI scans confirming measurable tumor size (lymph node must be >1cm in its longest transverse diameter). Measurement by physical exam is acceptable in the case of palpable and reproducibly measurable axillary or other superficial tumors.
4. Positive expression of cluster of differentiation antigen 20 (CD20) by biopsy or circulating lymphocytes.
5. Zero or one prior chemotherapeutic or immunotherapeutic treatment regimen for B-cell NHL.
6. Male or female greater than or equal to 18 years of age.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
8. Adequate renal function: Creatinine less than 1.5 mg/dL; blood urea nitrogen (BUN) less than 30 mg/dL or a creatinine clearance greater than or equal to 60 mL/min based on calculation of creatinine clearance using the Cockcroft-Gault method or from a 24-hour urine collection. Creatinine clearance 40- 59 mL/min from a 24-hour urine collection would require a Nipent dose reduction of 25%. Patients with a Creatinine clearance <40 mL/min from a 24-hour urine collection will be excluded.
9. Adequate bone marrow function: absolute neutrophil count (ANC) greater than or equal to 1,000 cells/µL; Platelet count greater than or equal to 75,000 cells/µL; Hemoglobin greater than or equal to 9 g/dL. Patients with idiopathic thrombocytopenia or autoimmune hemolytic anemia are eligible with prior approval of Sponsor Investigator.
10. Adequate liver function: Bilirubin less than or equal to 2.0 mg/dL; AST and ALT less than or equal to 5 times upper limit of normal (ULN).
11. Adequate cardiac function in the judgment of the Investigator, including New York Heart Association (NYHA) classification of I or II.
12. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration.
13. Patient agrees to use an acceptable method of birth control, if fertile patient (male or female), to avoid pregnancy for the duration of the study and for at least 3 months thereafter.
14. Completed Patient Informed Consent Form.

Exclusion Criteria:

1. Previous or current intermediate or high-grade lymphoma.
2. White blood cell count (WBC) greater than 30,000 cells/µL.
3. Received prior therapy using Rituxan, unless such therapy was completed at least 6 months prior to study registration. Patients whose disease was non-responsive to prior Rituxan therapy will be excluded.
4. Known sensitivity to Nipent, Rituxan, Cytoxan or any component of these drugs.
5. Patient received replacement steroid therapy less than 4 weeks prior to study registration.
6. History of other malignancy that could affect the diagnosis or assessment of the study treatment.
7. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) illness.
8. Known prior history of and/or active viral hepatitis (HBV or HCV).
9. Patient is unable to comply with the requirements of this study.
10. Patients with Richter's transformation will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Samaniego, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 29, 2005 to July 26, 2007. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 100 participants recruited, fifteen were excluded as screen failures prior to study assignment leaving an enrollment of 85 for the study.
Groups:
- Cytoxan + Rituxan + Nipent: Cytoxan 600 mg/m^2, Rituxan 375 mg/m^2 and Nipent 4 mg/m^2 on Day 1 of 21 Day Cycle.
Period: Overall Study
Arm/Group | Cytoxan + Rituxan + Nipent
Started | 85
Completed | 78
Not Completed | 7
Not completed — Ineligible | 2
Not completed — Death | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cytoxan + Rituxan + Nipent
Number analyzed (Participants) | 85
Age, Continuous [Median (Full Range); unit: years] | 59 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Participant Response Rate According to the International Working Group (IWG) Response Criteria for Non Hodgkin's Lymphoma (NHL), Cheson 1999
Description: Number of participants with response out of total treated participants using IWG defined 6 categories based on IWG 1999 Response Criteria for NHL of efficacy response or nonresponse to treatment in non-Hodgkins lymphoma (NHL): complete remission (CR), complete remission/unconfirmed (CRu), partial remission (PR), stable disease (SD). CR: is a complete disappearance of all disease with the exception of nodes. No new lesions. Previously enlarged organs must have regressed and not be palpable. Bone marrow(BM) must be negative if positive at baseline. Normalization of markers. CR Unconfirmed (CRU) does not qualify for CR above, due to a residual nodal mass or an indeterminate BM. PR: is a 50% decrease in the sum of the products of diameters (SPD) for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions. SD: participants who have achieved less than a PR but who have not developed findings consistent with progressive disease.
Time Frame: Evaluated after treatment in Cycles 3, 6 and 9 (1 Cycle = 21 Days), up to 7 months
Population: Two participants of the 85 enrolled were found to be ineligible following the enrollment and not treated therefore are excluded from outcome analysis. For the 83 eligible participants, five were considered inevaluable for response, but are included as non-responders in an intent-to-treat analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cytoxan + Rituxan + Nipent
Number analyzed (Participants) | 83
Percentage of Participants
  CR/CRu | 86.8
  Overall response | 91.6

2. Primary Outcome: Number of Participants With Complete Response (CR)/Complete Response Unconfirmed (CRu) With Low-grade Lymphoma (N=83) After 6-9 Cycles of PCR Therapy
Description: Number of participants with response according to the International Working Group (IWG) anatomic criteria for assessing six categories of efficacy response or nonresponse to treatment in non-Hodgkins lymphoma (NHL): complete remission (CR), complete remission/unconfirmed (CRu), partial remission (PR), stable disease (SD), relapsed disease (RD), and progressive disease (PD). Response was assessed after 3, 6, and 9 cycles of therapy.
Time Frame: 9 cycles of 21 days, up to 7 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cytoxan + Rituxan + Nipent
Number analyzed (Participants) | 83
participants | 72

3. Secondary Outcome: 3-Year Progression-Free Survival
Description: Progression-free survival (PFS) was defined as time from initiation of therapy to progression of disease or death, whichever occurred first. The Kaplan-Meier method was used to estimate PFS.
Time Frame: PFS assessed 7 days prior to every cycle and then every 3 months after off-treatment for one year, every 6 months for second year, then once on third year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cytoxan + Rituxan + Nipent
Number analyzed (Participants) | 83
percentage of participants | 73 [64 to 83]

ADVERSE EVENTS:
Time Frame: Adverse event reporting period begins upon first administration of study drug and continues until 30 calendar days after the last exposure to study drug. Treatment includes from one to nine 21-day cycles.
Arm/Group | Cytoxan + Rituxan + Nipent
Serious Adverse Events (participants affected / at risk) | 6/83
Other Adverse Events (participants affected / at risk) | 83/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytoxan + Rituxan + Nipent (N=83)
FATIGUE (General disorders) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytoxan + Rituxan + Nipent (N=83)
ALLERGIC REACTION (Immune system disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 5 (5)
AUDITORY/ EAR (OTHER) (Ear and labyrinth disorders) | 1 (1)
BLURRED VISION (Eye disorders) | 13 (13)
CONSTIPATION (Gastrointestinal disorders) | 29 (29)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 38 (38)
DIZZINESS (Psychiatric disorders) | 18 (18)
DRY EYE (Eye disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 21 (21)
EDEMA, FACIAL (General disorders) | 11 (11)
EDEMA, LIMB (General disorders) | 12 (12)
FATIGUE (General disorders) | 65 (65)
FEVER NEUTROPENIC (Infections and infestations) | 1 (1)
FEVER WITHOUT NEUTROPENIA (Infections and infestations) | 30 (30)
NOSE BLEED (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INDIGESTION (Gastrointestinal disorders) | 1 (1)
INFECTION WITH NORMA ANC (Infections and infestations) | 11 (11)
INSOMNIA (General disorders) | 1 (1)
MEMORY IMPAIRMENT (Psychiatric disorders) | 9 (9)
MOOD ALTERATION (Psychiatric disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 49 (49)
NAUSEA (Gastrointestinal disorders) | 67 (67)
NEUROPATHY, SENSORY (Nervous system disorders) | 17 (17)
PAIN (BACK) (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN (BONE) (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN (CHEST/THORAX) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN (DENTAL/ TEETH) (Gastrointestinal disorders) | 1 (1)
PAIN (HEADACHE) (Nervous system disorders) | 10 (10)
PAIN (MIDDLE EAR) (Ear and labyrinth disorders) | 1 (1)
PAIN (ORAL CAVITY) (Gastrointestinal disorders) | 20 (20)
PAIN (OTHER) (General disorders) | 1 (1)
PAIN (STOMACH) (Gastrointestinal disorders) | 1 (1)
PRURITUS/ ITCHING (Skin and subcutaneous tissue disorders) | 4 (4)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 5 (5)
REDNESS OF EYES (Eye disorders) | 26 (26)
RIGORS/ CHILLS (General disorders) | 2 (2)
SENSORY (Nervous system disorders) | 5 (5)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SWEATING (Skin and subcutaneous tissue disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 45 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes